CLINICAL TRIAL: NCT04657809
Title: "Insulin Fast Dissolving Film for Intranasal Delivery Via Olfactory Region, a Promising Approach for the Treatment of Anosmia in COVID 19 Patients: Design, In-vitro Characterization and Clinical Evaluation."
Brief Title: Clinical Assessment of Insulin Fast Dissolving Film in Treatment of Post Infection Anosmia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soad Ali (Other)
Collaborators: Minia University (Other)
Responsible Party: Sponsor-Investigator, Soad Ali, Assistant Professor, Deraya University
Organization: Deraya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S85insu23fdf
Record Dates: First submitted 2020-12-02; First posted 2020-12-08 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin fast dissolving film (Experimental): Formulated bioadhesive fast dissolving film contains 100IU of insulin
  Interventions: Combination Product: Insulin film; Device: Fast dissolving film
- Plain fast dissolving film (Placebo Comparator): Formulated bioadhesive fast dissolving film contains no drug
  Interventions: Combination Product: Insulin film; Device: Fast dissolving film

INTERVENTIONS:
Combination Product: Insulin film — Insulin suspension vials
Device: Fast dissolving film — Fast dissolving film

SUMMARY:
The study aimed to investigate the efficacy of insulin in a new dosage form ( fast dissolving film) in treatment of anosmia in patients post infested with Covid-19. The study implication based in two methods evaluations

1. Threshold test
2. identification test.

DETAILED DESCRIPTION:
This study was designed to improve smell disorders after corona infection that is very anxious for all patients.

Inclusion criteria were loss of smell, post covid-19 infection, age from 18 to 70 years and accept sharing and follow up.

The application of dosage form by ENT specialist at otorhinolaryngology clinic at Minia University hospital. Dose was 100iu of insulin 3 times weekly for 4 weeks. The new dosage form with insulin was compared with a placebo to ensure statistical improvement.

The tests were performed in each visit. Primary outcome was the improvement of smell sensors in those patients

ELIGIBILITY:
Inclusion Criteria:

* anosmia post covid-19 infection

Exclusion Criteria:

* nasal polyps or fractions or syrgery in nose from 6 months or less

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Smell sensation improvement | 4 weeks
  By decrease the threshold sensation with butanol test

CONTACTS AND LOCATIONS:
Overall Officials: Soad Mohamed, Study Director — Deraya
Locations (1):
- Soad, Minya, Egypt

REFERENCES:
- [Derived] Webster KE, O'Byrne L, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the prevention of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013877. doi: 10.1002/14651858.CD013877.pub3. PMID 36063364
- [Derived] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013876. doi: 10.1002/14651858.CD013876.pub3. PMID 36062970